CLINICAL TRIAL: NCT00475020
Title: Allogeneic Stem Cell Transplantation for Myelofibrosis and Myelodysplastic Syndrome Using Reduced Intensity Busulfan and Fludarabine Conditioning
Brief Title: Allogeneic Stem Cell Transplantation for Myelofibrosis and Myelodysplastic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0726; NCI-2012-01477 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2007-05-15; First posted 2007-05-17 (Estimated); Results first posted 2018-12-04 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Myelofibrosis
Keywords: Idiopathic Myelofibrosis; Myelofibrosis; Essential Thrombocythemia; Polycythemia Vera; Busulfan; Antithymocyte Globulin; ATG; Fludarabine; Thymoglobulin
MeSH Terms: conditions — Primary Myelofibrosis; Thrombocythemia, Essential; Polycythemia Vera | interventions — Busulfan; fludarabine; fludarabine phosphate; thymoglobulin; Antilymphocyte Serum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Fludarabine + Busulfan + Thymoglobulin (Experimental): Fludarabine 40 mg/m^2 by vein daily over 1 hour x 4 days. Busulfan test dose = 32 mg/m^2 by vein x 1 day; 100 mg/m^2 by vein daily over 3 hours x 4 days. Thymoglobulin 2.5 mg/kg by vein over 6 hours x 3 days if there is an unrelated or a mismatched donor.
  Interventions: Drug: Busulfan; Drug: Fludarabine; Drug: Thymoglobulin (ATG)

INTERVENTIONS:
Drug: Busulfan — Test dose = 32 mg/m^2 by vein x 1 day; 100 mg/m^2 by vein daily over 3 hours x 4 days
  Other Names: Busulfex; Myleran
Drug: Fludarabine — 40 mg/m^2 by vein daily over 1 hour x 4 days
  Other Names: Fludarabine Phosphate
Drug: Thymoglobulin (ATG) — 2.5 mg/kg by vein over 6 hours x 3 days if there is an unrelated or a mismatched donor
  Other Names: Antithymocyte Globulin; Thymoglobulin; ATG

SUMMARY:
The goal of this clinical research study is to learn if using a combination of fludarabine, busulfan, and antithymocyte globulin (ATG) can help to control myelofibrosis or myelodysplastic syndrome in patients receiving a bone marrow or blood stem cell transplant. The safety of these drugs will also be studied.

DETAILED DESCRIPTION:
Busulfan is a chemotherapy drug that kills cancer cells by binding to DNA, and is commonly used in stem cell transplants. Fludarabine is a drug that has anti-leukemia and immunosuppressive effects. ATG helps to reduce the risk of transplant rejection and to prevent graft versus host disease.

You will receive fludarabine by vein over 1 hour on Days -5 to -2. You will receive busulfan by vein over 3 hours on Day -5 to -2 immediately after completing fludarabine. If you have an unrelated or a mismatched donor, you will receive ATG by vein over 6 hours on Days -3 to -1 to prevent graft versus host disease and to help engraftment.

You will first receive a low-level "test" dose of busulfan, and blood samples (about 1 teaspoon each time) will be drawn for pharmacokinetic (PK) tests. This may be done as an outpatient prior to inpatient admission. PK tests measure the level of the study drug in the blood over different time points. This information will be used to decide the next dose needed to reach the target blood level that matches your body size.

About 11 total samples of blood will be drawn for PK testing after the test dose and before the first high-dose busulfan treatment. A heparin lock will be placed in your vein to lower the number of needle sticks needed for these draws. If it is not possible for these blood level tests to be performed for technical or scheduling reasons or for any other reason, you will receive the standard fixed busulfan dose without the "test dose."

You will receive the donor bone marrow or blood stem cells by vein over about 1 hour on Day 0.

Two (2) days before the stem cell infusion on Day -2, tacrolimus will be started as a non-stop infusion by vein and will be changed to oral tablets before you leave the hospital. You will continue to take tacrolimus by mouth, for at least 4 months.

Four (4) doses of Methotrexate will be give as a short infusion Day 1, Day 3, Day 6 and Day 11 after stem cell infusion. Both these are given to decrease the risk of getting graft-vs-host disease (GvHD). Further immunosuppressive therapy with methylprednisolone (a steroid) or other drugs may also be used to treat GvHD if it occurs.

You will have 3 teaspoonfuls of blood drawn for routine tests every day while you are in the hospital and at least 2 times a week for the first 100 days after transplant. You may need frequent blood transfusions and may have to be admitted to the hospital to receive antibiotics if you get a fever. Three (3) teaspoonful of blood and a bone marrow aspirate and biopsy will be taken 1 month, 3 months, 6 months, 12 months, 18 months, and 24 months after the transplant to check the response to the treatment. After the first 2 years, your disease status will be followed by a yearly phone call or letter from you or your regular doctor to the study doctor.

Tests and/or procedures may be performed before the scheduled time, if your doctor thinks it is needed.

You will be taken off the study if your disease gets worse or if further treatment is not in your best interest.

This is an investigational study. All the drugs to be used in this study are FDA approved and commercially available. About 110 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Idiopathic Myelofibrosis or Myelofibrosis secondary to Polycythemia Vera or Essential Thrombocythemia or Myelodysplastic syndrome with or without fibrosis.
2. Patients 75 years or younger
3. Patients must have an HLA matched or at least a 9/10 antigen (A, B, C, DQ or DR) matched related or unrelated donor.
4. Patients must have a Zubrod PS 2 or less.
5. Creatinine < 1.6 mg/dl
6. Ejection fraction >/= 40%, unless cleared by cardiology
7. Serum direct bilirubin < 2 mg/dl (unless due to Gilbert's syndrome), serum glutamate pyruvate transaminase (SGPT) </= 4 x normal values
8. Forced expiratory volume at one second (FEV1), forced vital capacity (FVC), or diffusing capacity of lung for carbon monoxide (DLCO) >/= 40% of expected.
9. Negative Beta human chorionic gonadotropin (HCG) test in a woman with child bearing potential defined as not post-menopausal for 12 months or no previous surgical sterilization.

Exclusion Criteria:

1. Uncontrolled life-threatening infections
2. HIV positive
3. Patients with Active viral hepatitis

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2006-01-04 (Actual); Primary Completion 2017-10-04 (Actual); Study Completion 2017-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Uday Popat, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants With Myelofibrosis and Myelodysplastic Syndrome: Allogeneic stem cell transplantation (SCT) with preparative regimen of fludarabine and busulfan in myelofibrosis and myelodysplastic syndrome
Period: Overall Study
Arm/Group | Participants With Myelofibrosis and Myelodysplastic Syndrome
Started | 63
Completed | 58
Not Completed | 5
Not completed — Physician Decision | 3
Not completed — Insurance Denial | 1
Not completed — Donor not able to donate the last minute | 1

BASELINE CHARACTERISTICS:
Arm/Group | Participants With Myelofibrosis and Myelodysplastic Syndrome
Number analyzed (Participants) | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 45
  >=65 years | 13
Age, Continuous [Median (Full Range); unit: years] | 59 [27 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 53
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 58

OUTCOME MEASURES:

1. Primary Outcome: Rate of Non-relapse Mortality at 100 Days Post-transplant
Description: To evaluate the safety of Fludarabine/Busulfan as conditioned regimen for allogeneic stem cell transplantation in patients with myelofibrosis/myelodysplastic syndrome at 100 days post-transplant
Time Frame: Non-relapse mortality at 100 days post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Myelofibrosis and Myelodysplastic Syndrome
Number analyzed (Participants) | 58
Participants
  Infections | 1
  Organ Failures | 2
  Sudden death: likely due to ischemic cardiac event | 1

2. Secondary Outcome: Efficacy of This Therapy 3 Years Post-transplant
Description: Efficacy Assessed as Number of Participants with Overall Survival, Leukemia Progression, Primary Graft Failure and Complete Hematological Response. Primary graft failure is defined as failure to achieve an ANC >/= 0.5 x 10 (9)/L for 3 consecutive days and evidence of donor chimerism by Day +28. Complete hematological response is defined by hemoglobin >/= 120 g/L; or achievement of transfusion independence, with stable Hb > 110 g/L, for RBC transfusion-dependent participants; Spleen not palpable; platelet count 150 x 10 (9)/L; White blood cell 4 x 10 (9)/L to 10 x 10(9)/L.
Time Frame: Up to 3 years post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Myelofibrosis and Myelodysplastic Syndrome
Number analyzed (Participants) | 58
Participants
  Overall survival at 3 years | 25
  Leukemia progression | 27
  Primary graft failures | 0
  Complete hematological remission | 44

ADVERSE EVENTS:
Time Frame: January 2006 to May 2012
Arm/Group | Participants With Myelofibrosis and Myelodysplastic Syndrome
All-Cause Mortality (participants affected / at risk) | 8/58
Serious Adverse Events (participants affected / at risk) | 18/58
Other Adverse Events (participants affected / at risk) | 58/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Myelofibrosis and Myelodysplastic Syndrome (N=58)
GI GvHD (Gastrointestinal disorders) | 2
Skin GvHD (Skin and subcutaneous tissue disorders) | 1
Infectious pneumonia (Infections and infestations) | 3
Veno-occlusive disease (Hepatobiliary disorders) | 2
Liver GvHD (Blood and lymphatic system disorders) | 1
Secondary graft failure (Blood and lymphatic system disorders) | 6
Hemolytic anemia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Renal failure (Renal and urinary disorders) | 2
Elevated transminitis (Hepatobiliary disorders) | 6
Septic shock (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Myelofibrosis and Myelodysplastic Syndrome (N=58)
Infections (Infections and infestations) | 34
Poor graft function (Blood and lymphatic system disorders) | 1
ABO incompatibility (Blood and lymphatic system disorders) | 1
ATG induced fevers (Investigations) | 24
Fluid overload (Investigations) | 22
GI GvHD (Gastrointestinal disorders) | 6
Mucositis (Gastrointestinal disorders) | 43
Upper GI GvHD (Gastrointestinal disorders) | 11
Renal insufficiency (Renal and urinary disorders) | 8
Liver GvHD (Hepatobiliary disorders) | 5
Veno-occlusive disease (Hepatobiliary disorders) | 1
Neutropenic fevers (Investigations) | 14
Headaches (General disorders) | 5
Infectious pneumonia (Infections and infestations) | 9
ATG induced shortness of breath (Respiratory, thoracic and mediastinal disorders) | 2
Skin GvHD (Skin and subcutaneous tissue disorders) | 14
Hypertension (Cardiac disorders) | 3
Ascites (Hepatobiliary disorders) | 2
Diarrhea (Gastrointestinal disorders) | 11
Hemorrhagic cystits (Renal and urinary disorders) | 2
Nausea (Gastrointestinal disorders) | 51
BK virus associated hemorrhagic cystitis (Infections and infestations) | 5
Elevated transminitis (Hepatobiliary disorders) | 20
Altered mental status changes (Nervous system disorders) | 3
Cytokine release syndrome (Investigations) | 2
Cellulitis (Skin and subcutaneous tissue disorders) | 2
ATG induced skin rash (Skin and subcutaneous tissue disorders) | 1
Fevers (Investigations) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-03-09): https://cdn.clinicaltrials.gov/large-docs/20/NCT00475020/Prot_SAP_000.pdf